CLINICAL TRIAL: NCT05558670
Title: Assessing Brain Network Characteristics in Patients With Disorders of Consciousness by Simultaneous Trimodal Positron Emission Tomography-Functional Magnetic Resonance Imaging-Electroencephalograph（PET-fMRI-EEG）Imaging
Brief Title: Brain Network Characteristics in Patients With Disorders of Consciousness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20222068
Record Dates: First submitted 2022-09-01; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-08

CONDITIONS: Disorders of Consciousness
Keywords: PET-fMRI-EEG; brain network; coma; Vegetative state(VS); Unresponsive wakefulness syndrome (UWS); Minimally conscious state(MCS); Emerged from minimally conscious state(EMCS)
MeSH Terms: conditions — Consciousness Disorders; Coma; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- coma
  Interventions: Other: PET-fMRI-EEG
- VS/UWS
  Interventions: Other: PET-fMRI-EEG
- MCS
  Interventions: Other: PET-fMRI-EEG
- EMCS
  Interventions: Other: PET-fMRI-EEG

INTERVENTIONS:
Other: PET-fMRI-EEG — Participants perform PET, fMRI, and EEG simultaneously using a MRI compatible EEG cap

SUMMARY:
Simultaneous measurement of the three modalities, functional magnetic resonance imaging (fMRI), positron emission tomography (PET) and electroencephalography (EEG) was proven to be feasible and advantageous in evaluating brain structural and functional (via fMRI), metabolic (via PET) and electrophysiological (via EEG) signatures simultaneously under the same conditions. Investigators use trimodal PET-fMRI-EEG imaging to explore the characteristics of brain network damage in patients with disorders of consciousness(DOC), assess the trajectory of consciousness recovery in a prospective observational cohort study.

ELIGIBILITY:
Inclusion Criteria:

1. Coma, VS/UWS, MCS and EMCS according to diagnostic criteria
2. Age ≥18 years
3. Written informed consent obtained

Exclusion Criteria:

1. Patients with contraindications to PET, MRI, EEG examinations or inability to complete PET-fMRI-EEG examinations (presence of ferromagnetic metal implants or hyperthermia)
2. Hyperglycemia that is difficult to correct
3. Patients with long-term use of corticosteroids
4. Patients with coexisting severe systemic disease and limited life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are selected in patients hospitalised in neurology department of Xijing hospital
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
CRS-R total score | Patients in coma after 3 weeks enrolled
  The coma recovery scale-revised(CRS-R) total score is used to measure level of consciousness of disorder in enrolled patients. CRS-R consists of six subscales addressing auditory, visual, motor, verbal, communication, and arousal functions.The lowest item on each subscale represents reflexive activity and the highest item represents cognitively mediated behavior. Maximum scores of each subscale are summed to obtain the total score (from 0 to 23).The score for each subscale is based on the presence or absence of a specific behavioral response to a sensory stimulus (higher scores are better).
GOSE score | Patients are followed up for 6 months after enrolled
  Glasgow Outcome Scale-Extended(GOSE) score is used to measure the functional limitations of participants. GOSE is a 1-8 point scale (1 = Death, 2 = Vegetative State, 3 = Lower Severe Disability, 4 = Upper Severe Disability, 5 = Lower Moderate Disability, 6 = Upper Moderate Disability, 7 = Lower Good Recovery, and 8 = Upper Good Recovery). Patients with higher scores are more independent.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, Study Director — Xijing Hospital
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No